CLINICAL TRIAL: NCT03226340
Title: Evaluation of the Efficacy and Safety of S-amlodipine+Chlorthalidone Combination Therapy and S-amlodipine+Telmisartan Combination Therapy in Hypertensive Patients Inadequately Controlled With Calcium Channel Blocker Monotherapy
Brief Title: S-amlodipine+Chlorthalidone vs S-amlodipine+Telmisartan in Hypertension
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Bundang Hospital (Other)
Collaborators: Hanlim Pharm. Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Dong-Ju Choi, Professor, MD, PhD, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HL_LDN_504
Record Dates: First submitted 2017-07-17; First posted 2017-07-21 (Actual); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Essential Hypertension
MeSH Terms: conditions — Essential Hypertension | interventions — levamlodipine; Chlorthalidone; Telmisartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- S-amlodipine + Chlorthalidone (Experimental): patients will receive S-amlodipine 2.5mg + Chlorthalidone 25mg p.o. once a day for 12 weeks.
  Interventions: Drug: S-amlodipine 2.5mg + Chlorthalidone 25mg
- S-amlodipine + Telmisartan (Active Comparator): patients will receive S-amlodipine 2.5mg + Telmisartan 40mg p.o. once a day for 12 weeks.
  Interventions: Drug: S-amlodipine 2.5mg + Telmisartan 40mg

INTERVENTIONS:
Drug: S-amlodipine 2.5mg + Chlorthalidone 25mg — patients will receive S-amlodipine 2.5mg + Chlorthalidone 25mg p.o. once a day for 12 weeks.
  Arms: S-amlodipine + Chlorthalidone
Drug: S-amlodipine 2.5mg + Telmisartan 40mg — patients will receive S-amlodipine 2.5mg + Telmisartan 40mg p.o. once a day for 12 weeks.
  Arms: S-amlodipine + Telmisartan

SUMMARY:
Evaluation of the Efficacy and Safety of S-amlodipine+Chlorthalidone Combination Therapy and S-amlodipine+Telmisartan Combination Therapy in Hypertensive Patients Inadequately Controlled With CCB(Calcium Channel Blocker) Monotherapy

DETAILED DESCRIPTION:
The aim of this study is to verify the difference at week 12 from the baseline value in the average variation of diastolic blood pressure (sitDBP) of the study group in which S-amlodipine / Chlorthalidone combination therapy is to be used in patients with essential hypertension who did not adequately respond to monotherapy of amlodipine or S-amlodipine, compared to the control group, in which a combination therapy of S-amlodipine / telmisartan is to be used.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women with essential hypertension who were aged 19 years or older and younger than 80 years
2. Patients who have been treated with amlodipine or S-amlodipine monotherapy for more than 2 weeks immediately before visit 1 (screening)
3. Visit 1 (screening) reference mean blood pressure measured three times in the arm is greater than sit DBP 90 mmHg
4. Those who have voluntarily agreed in writing to participate in the trial

Exclusion Criteria:

1. Patients with a history of secondary hypertension and all those with suspected secondary hypertension (including, but not limited to, coarctation of the aorta, primary aldosteronism, renal artery stenosis, Cushing's syndrome, chromium-rich cell tumor, polycystic kidney disease, etc.)
2. Patients with a mean SBP of 200 mmHg or more or a sit DBP of 110 mmHg or more at visit 1.
3. When the blood pressure was measured three times in the reference arm of visit 1 (screening), the difference between the highest lowest sit SBP was 20 mmHg or higher and the difference between the highest lowest sit DBP was 10 mmHg or higher.
4. An uncontrolled diabetic patient(HbA1c≥9.0%)
5. In addition to antihypertensive drugs, drugs that may affect blood pressure( Systemic steroids, Thyroid hormones, Oral contraceptives, antipsychotic drugs, NSAIDs, sympathomimetics, immunosuppressants, etc.) have been continuously administered for more than 12 weeks prior to visit 1 (screening)
6. Patients who are expected to take antihypertensive drugs other than clinical drugs during the trial
7. Patients with orthostatic hypotension with symptoms
8. Patients with a history of malignant tumors including leukemia and lymphoma within the past 5 years
9. Patients with a history of autoimmune diseases such as chronic joint rheumatism and systemic lupus erythematosus
10. Those who have a history of hypersensitivity to the amlodipine nicotinate or other chlortalidone or telmisartan drug
11. Patients with clinically significant renal • hepatic disease such as those on dialysis, cirrhosis, biliary obstruction, hepatic failure, or those who have the following findings on visit 1 (screening)

    * ALanine Transaminase or ASpartate Transaminase is more than 3 times the normal upper limit
    * Total bilirubin more than twice the normal upper limit
    * More than twice the Blood Urea Nitrogen normal upper limit
    * Alkaline Phosphatase More than twice the normal upper limit - Creatinine Clearance Less than 10 mL / min
12. Within the last 6 months, patients who have received the following diseases or treatments and whose clinical judgment is meaningful to the researcher

    * Severe heart disease (heart failure New York Heart Association class III and IV), ischemic heart disease, peripheral vascular disease, hemodynamically significant valve stenosis, arrhythmia, etc
    * Patients with severe cerebrovascular disorders (stroke, cerebral infarction, cerebral hemorrhage, etc.)
13. Shock patient
14. Patients with clinical history of alcohol or substance abuse
15. Patients with potential pregnancy or breastfeeding

    * In the case of pregnant women, if the negative is not confirmed during pregnancy test
    * Women who did not consent to contraception in a medically acceptable way during the trial
    * Medically acceptable contraceptive methods: use condoms, injectable or injectable contraceptives, intrauterine contraceptive device, etc.
16. If the tester judges that the participation in the clinical trial is not legal or mental character
17. Clinical studies with other clinical trial drugs within 4 weeks prior to screening patients with experience

Ages: 19 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2015-12-02 (Actual); Primary Completion 2018-03-31 (Estimated); Study Completion 2018-03-31 (Estimated)

PRIMARY OUTCOMES:
sit diastolic blood pressure | 12 weeks
  Mean change in sit diastolic blood pressure after 12 weeks compared to baseline.

SECONDARY OUTCOMES:
sit diastolic blood pressure | 6 weeks
  Mean change in sit diastolic blood pressure after 6 weeks compared to baseline.
sit systolic blood pressure | 12 weeks
  Mean change in sit systolic blood pressure after 6 weeks and 12 weeks compared to baseline.
Blood pressure normalization | 12 weeks
  Blood pressure normalization ratio after 12 weeks compared to baseline( sit systolic blood pressure <140 mmHg or sit diastolic blood pressure <90 mmHg).

CONTACTS AND LOCATIONS:
Locations (10):
- South Korea (10):
  - Hallym University Medical Center, Anyang, Dongan-gu
  - Kyung Hee University Hospital, Seoul, Dongdaemun-gu
  - Hallym University Medical Center, Seoul, Gangdong-gu,
  - Samsung Medical Center, Seoul, Gangnam-Gu
  - Korea Univ. Guro Hospital, Seoul, Guro
  - Seoul National University Hospital, Seoul, Jongno-gu
  - Hanyang University Medical Center, Seoul, Seongdong-gu
  - Asan Medical Center, Seoul, Songpa-gu
  - Ajou Univ. Medical Center, Suwon, Yeong-tong
  - Seoul National University Bundang Hospital, Seongnam

REFERENCES:
- [Derived] Jo SH, Park SJ, Kim EJ, Kim SJ, Cho HJ, Song JM, Shin J, Park JJ, Shin JH, Han KR, Choi DJ. S-amlodipine plus chlorthalidone vs. S-amlodipine plus telmisartan in hypertensive patients unresponsive to amlodipine monotherapy: study protocol for a randomized controlled trial. Trials. 2018 Jun 20;19(1):324. doi: 10.1186/s13063-018-2636-1. PMID 29925421